CLINICAL TRIAL: NCT05807503
Title: Evaluation of the Effect of Early Administered Neuroprotective Drug on Treatment Result in Patients After Traumatic Brain Injury - PILOT Trial
Brief Title: Evaluation of the Effect of Neuroprotective Drug on Treatment Result in Patients After Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Klaudyna Kojder, PhD, Pomeranian Medical University Szczecin
Other Study IDs: 02/10/2020
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: TBI; neuroprotective treatment; Cerebrolysin; neuromonitoring; NIRS; ICP; ONDS
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — cerebrolysin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A with Cerebrolysin administration: Group of patients with TBI diagnosis, admitted to ICU for further treatment after or without neurosurgical craniotomy, treated with Cerebrolysin administration in addition to standard ICU protocols.
  Interventions: Drug: Cerebrolysin
- B without Cerebrolysin administration: Group of patients with TBI diagnosis, admitted to ICU for further treatment after or without neurosurgical craniotomy, treated without Cerebrolysin administration according to standard ICU protocols.

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin administration in short period of time after TBI
  Groups: A with Cerebrolysin administration

SUMMARY:
Traumatic Brain Injury TBI is one of the most common causes of death and recovery failure worldwide. Each element of treatment, starting from possible surgical treatment, patient monitoring and neuroprotective treatment, can be important in the overall outcome of patients' treatment. More and more elements of treatment are discussed in the literature in the multimodal approach to the patient with a trauma to the central nervous system. Cerebrolysin is a drug with a proven beneficial effect on the prognosis of patients with TBI. In our trial we stated the hypothesis that Cerebrolysin in combination with multimodal monitoring and surgical craniotomy is beneficial for the patients. In retrospective analysis we divided the patients into two groups : with and without cerebrolysin. We also analyzed how cerebrolysin influences the treatment results with the combination with additional neuromonitoring of both invasive intracranial pressure (ICP) measurement and non-invasive saturation in the jugular vein, nirs, ultrasound of the optic nerve diameter. We also analyzed if there is any change in the results of treatment after combining Cerebrolysin with another neuroprotective drug : amantadine. We also analyzed the influence of craniotomy combined with cerebrolysin treatment. In an observational study, we collected information on 56 patients.

ELIGIBILITY:
Inclusion Criteria:

* TBI diagnosis
* admission to ICU
* age >18 y

Exclusion Criteria:

* initially lethal injury
* age <18 y

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 56 patients in age from 28 to 91 years old, 33% female, 66% male, bleeding during the TBI:
  * epidural: 16/56 (27%)
  * subdural : 26/56 (45%)
  * into deep structures: 14/56 (23%)
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale GOS | 2 months
  Glasgow Outcome Scale
Length Of Stay LOS | 2 months
  Length Of Stay
Mortality | 2 months
  Death of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Jarosz, Principal Investigator — The Department Of Specialist Nursing, Pomeranian Medical University
Locations (1):
- Pomeranian Medical University, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
more information after individual contacting with investigators